CLINICAL TRIAL: NCT00616889
Title: Effects of Seroquel on Sleep Architecture in Patients With Bipolar Depression or Major Depressive Disorder - An Open Label Study
Brief Title: Effect of Quetiapine on Sleep Architecture in Bipolar Depression and Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Principal Investigator, Queen's University
Other Study IDs: PSIY-206-05; D1449C00011
Record Dates: First submitted 2005-09-09; First posted 2008-02-15 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Seroquel added to medication regime and sleep quality measured
  Interventions: Drug: Seroquel

INTERVENTIONS:
Drug: Seroquel — The dosage is flexible from 50-600 mg based on the investigator's clinical judgement and patient tolerance. It may be raised or lowered at will.
  Other Names: Quetiapine

SUMMARY:
Clinical practice indicates that Quetiapine has sedating properties, and its sedative effects may play an important role in restoring quality of sleep in patients with various psychiatric conditions who frequently experience sleep disturbances as part of their illness. It is well known that depressive disorders are very frequently associated with significant sleep disturbance. Sleep disruption is a feature of Bipolar Disorder during both Depressed and Manic/Hypomanic episodes. Considering that Seroquel has good antidepressant properties (Calabrese, 2004), the investigators suggest that Seroquel's effect on sleep architecture contributes to its antidepressant properties.

DETAILED DESCRIPTION:
Primary Objective:

To assess the objective (polysomnographic) change in sleep quality before and after introduction of Seroquel (Quetiapine) in treatment of patients with Bipolar Depression or Major Depressive Disorder.

Secondary Objectives:

To assess the objective (polysomnographic) and subjective changes in sleep quality parameters before and at different stages after introduction of Seroquel (Quetiapine) treatment, longitudinally, and to correlate these changes with measures of illness severity.

Study Design:

Prospective polysomnographic (PSG) study of patients before and after treatment with Seroquel (Quetiapine). PSG recordings will be done three (optional four) times during the study: before starting the Seroquel (Quetiapine) (baseline), at day 2 to 4 (early) and day 21 to 28 (longer term). (Optional fourth PSG can be done at day 42-56). PSG will be completed at patients home with a portable PSG.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent;
2. A diagnosis of Bipolar Disorder Type 1,2 or NOS by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV);OR Major Depressive Disorder
3. Males or Females aged 18 years or more;
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment;
5. Able to understand and comply with the requirements of the study;
6. Current depressive episode with a HAM-D17 score of 15 or more.

Exclusion Criteria:

1. Current Manic, Hypomanic or Mixed episode, with YMRS 12 or more;
2. Current or past diagnosis of Schizophrenia;
3. Pregnant women, or women in childbearing age, not willing to use appropriate contraception or women currently nursing;
4. Patient on antipsychotic medication;
5. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others;
6. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator;
7. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir;
8. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids;
9. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization;
10. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria;
11. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen dependence by DSM-IV criteria within 4 weeks prior to enrolment;
12. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment;
13. Unstable or inadequately treated medical illness (e.g., diabetes, angina pectoris, hypertension) as judged by the investigator;
14. Involvement in the planning and conduct of the study;
15. Previous enrolment in the present study;
16. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements;
17. If participant's liver function testing is rated 2 in the upper limits of normal.
18. Diagnosis of Dementia
19. Regular use of benzodiazepines unless at a stable dose for at least 12 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with current Major Depressive Disorder or Bipolar Depression
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Sleep quality as measured by overnight PSG. | baseline, day 2 to 4 (early) and day 21 to 28 (longer term). Optional reading at day 42-56

CONTACTS AND LOCATIONS:
Overall Officials: Roumen V Milev, MD, Principal Investigator — Queen's University
Locations (1):
- Pccc, Mhs, Kingston, Ontario, Canada